CLINICAL TRIAL: NCT00506077
Title: A Phase IIa, Randomized, Double-Blind, Placebo-Controlled, 2-Period, Cross-Over Clinical Trial to Study the Safety and Efficacy of MK0249 for the Treatment of Cognitive Impairment in Patients With Schizophrenia
Brief Title: MK0249 for the Treatment of Cognitive Impairment in Patients With Schizophrenia (0249-016)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0249-016; 2007_522
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Results first posted 2011-03-07 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Paranoid Schizophrenia
Keywords: Undifferentiated schizophrenia; residual schizophrenia
MeSH Terms: conditions — Schizophrenia, Paranoid | interventions — MK-0249

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- MK0249 (Experimental)
  Interventions: Drug: MK0249
- Placebo (Placebo Comparator)
  Interventions: Drug: Comparator: Placebo (unspecified)

INTERVENTIONS:
Drug: MK0249 — MK0249 10mg (2 x 5 mg) tablet daily (qd) for 28 days.
  Arms: MK0249
Drug: Comparator: Placebo (unspecified) — MK0249 10mg (2 x 5 mg) Pbo tablet qd for a 28 day treatment period.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of an investigational drug MK0249 for the treatment of the cognitive impairment in patients with schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Patient is clinically stable, on current antipsychotic medication for at least 3 months and current dose for 2 months
* Patient has a 6th grade reading level or better
* Females are not pregnant, and those who can have children agree to remain abstinent or use acceptable birth control throughout the study
* Patient has had a stable living arrangement for at least 3 months prior to study start
* Patient is in general good health based on screening assessments
* Patient has total Positive and Negative Syndrome Scale (PANSS) score between 36 and 75 at screening and at the first baseline visit
* Patient has a Clinical Global Impressions - Severity (CGI-S) score less than or equal to 4 at screening and at the first baseline visit

Exclusion Criteria:

* Patient has a major disease/disorder that may interfere with cognitive testing (such as mental retardation) and/or pose a risk upon study participation
* Patient has a history of head trauma with loss of consciousness greater than 15 minutes
* Patient has had warfarin treatment, MAO inhibitors, clonazepam or clozapine within 1 month of screening
* Patient has had ECT treatment within 6 months of screening
* Patient requires treatment with antihistamines or certain other medications listed in the protocol
* Patient has a history of liver disease that has been active within the last 2 years, or a history of cancer within the past 5 years
* Patient has a history of alcohol or drug dependence within the past year or alcohol or drug abuse within 3 months of screening

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2007-12; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Derived] F Egan M, Zhao X, Gottwald R, Harper-Mozley L, Zhang Y, Snavely D, Lines C, Michelson D. Randomized crossover study of the histamine H3 inverse agonist MK-0249 for the treatment of cognitive impairment in patients with schizophrenia. Schizophr Res. 2013 May;146(1-3):224-30. doi: 10.1016/j.schres.2013.02.030. Epub 2013 Mar 22. PMID 23523692

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient Dosed: 11 February 2008; Last Patient Last Treatment: 08 October 2008. Six ex-U.S. study centers (3 Russia, 3 India).
Pre-assignment Details: At visit 1, patients were assessed using the protocol eligibility criteria. Eligible patients continued into an 8 day single-blind placebo washout/run-in period, and then were randomized at visit 3 to 1 of 2 cross-over treatment sequences.
Groups:
- MK0249 Then Placebo: These subjects received MK0249 during Treatment Period 1 and Placebo during Treatment Period 2.
- Placebo Then MK0249: These subjects received Placebo during Treatment Period 1 and MK0249 during Treatment Period 2.
Period: Treatment Period 1
Arm/Group | MK0249 Then Placebo | Placebo Then MK0249
Started | 28 | 27
Completed | 24 | 24
Not Completed | 4 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 2 | 0
Period: Washout
Arm/Group | MK0249 Then Placebo | Placebo Then MK0249
Started | 24 | 24
Completed | 24 | 24
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | MK0249 Then Placebo | Placebo Then MK0249
Started | 24 | 24
Completed | 23 | 23
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK0249 Then Placebo | Placebo Then MK0249 | Total
Number analyzed (Participants) | 28 | 27 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.7 (7.5) | 32.5 (8.4) | 31.6 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at 4 Weeks of Treatment in Total Cognitive Score on the Brief Assessment of Cognition in Schizophrenia (BACS) Battery.
Description: The mean change from baseline after 4 weeks of treatment in total cognitive score on the BACS was calculated as a weighted average of T-scores (normalized for age) from BACS subtests including Verbal Memory, Digit Sequencing, Token Motor, Symbol Coding, Semantic Fluency, Letter Fluency, and Tower of London. The minimum and maximum values possible for this composite T-score of the change from baseline were -131 and 131, respectively. Higher values (positive changes from baseline) indicate better performance.
Time Frame: Baseline and 4 weeks of treatment
Population: Full Analysis Set (FAS): The FAS included all randomized patients who took at lease one dose of study medication and had at least one post-randomization efficacy measurement in either of the two treatment periods. The data as observed (DAO) approach was used to handle missing data.
Measure: Least Squares Mean (95% Confidence Interval); unit: Composite T-score
Groups:
- MK0249: 10 mg per day of MK-0249 were taken orally for Treatment Period 1 or Treatment Period 2 (depending on the sequence). At any time after 3 days of double-blind treatment if patients who were unable to tolerate 10 mg per day, they were allowed to titrate down to 7 mg per day and remained on 7 mg per day for the remainder of the treatment period.
- Placebo: 10 mg per day of matching placebo were taken orally for Treatment Period 1 or Treatment Period 2 (depending on the sequence). At any time after 3 days of double-blind treatment if patients who were unable to tolerate 10 mg per day, they were allowed to titrate down to 7 mg per day and remained on 7 mg per day for the remainder of the treatment period.
Arm/Group | MK0249 | Placebo
Number analyzed (Participants) | 47 | 46
Composite T-score | 0.4 [-1.2 to 2.1] | 0.5 [-1.1 to 2.2]
Statistical Analysis 1: Comparison: MK0249 vs Placebo; Test type: Superiority or Other; p = 0.939, constrained longitudinal data analysis — The Benjamini & Hochberg False Discovery Rate (FDR) approach at critical value 0.05 was used among 1 primary and 3 secondary cognition efficacy endpoints to control the false positive rate; The model factors were treatment, sequence, period, week (as categorical variable), site, treatment-by-week, sequence-by-week, and period-by-week

2. Secondary Outcome: Mean Change From Baseline at 4 Weeks of Treatment in Attention/Processing Speed Composite Score
Description: The Attention/Processing Speed Composite Score was comprised of the University of Pennsylvania's Computerized Neuropsychological Battery (CNP) Penn Continuous Performance Test (PCPT) and BACS battery Symbol Coding. The composite score was calculated as a weighted average of the T-scores (normalized for age) for each test. The minimum and maximum values possible for this composite T-score of the change from baseline were -91 and 91, respectively. Higher values (positive changes from baseline) indicate better performance.
Time Frame: Baseline and 4 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Composite T-score
Arm/Group | MK0249 | Placebo
Number analyzed (Participants) | 45 | 45
Composite T-score | 0.5 [-0.4 to 1.5] | 0.0 [-0.9 to 0.9]
Statistical Analysis 1: Comparison: MK0249 vs Placebo; Test type: Superiority or Other; p = 0.736, constrained Longitudinal Data Analysis — P-Value Comments (limit 250 characters): The Benjamini & Hochberg False Discovery Rate (FDR) approach at critical value 0.05 was used among 1 primary and 3 secondary cognition efficacy endpoints to control the false positive rate; [statistical method as in outcome 1, analysis 1]

3. Secondary Outcome: Mean Change From Baseline at 4 Weeks of Treatment in Episodic Memory Composite Score
Description: The Episodic Memory Composite Score was comprised of the University of Pennsylvania's Computerized Neuropsychological Battery (CNP) Face Memory and BACS battery Verbal Memory. The composite score was calculated as a weighted average of the T-scores (normalized for age) for each test. The minimum and maximum values possible for this composite T-score of the change from baseline were -202 and 202, respectively. Higher values (positive changes from baseline) indicate better performance.
Time Frame: Baseline and 4 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Composite T-score
Arm/Group | MK0249 | Placebo
Number analyzed (Participants) | 47 | 45
Composite T-score | 0.9 [-0.9 to 2.6] | 0.1 [-1.6 to 1.8]
Statistical Analysis 1: Comparison: MK0249 vs Placebo; Test type: Superiority or Other; p = 0.736, constrained Longitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

4. Secondary Outcome: Mean Change From Baseline at 4 Weeks of Treatment in Working Memory Composite Score
Description: The Working Memory Composite Score was comprised of the University of Pennsylvania's Computerized Neuropsychological (CNP) battery N-back test and the BACS battery Digit Sequencing test. The composite score was calculated as a weighted average of the T-scores (normalized for age) for each test. The minimum and maximum values possible for this composite T-score of the change from baseline were -122 and 122, respectively. Higher values (positive changes from baseline) indicate better performance.
Time Frame: Baseline and 4 weeks of treatment
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Composite T-score
Arm/Group | MK0249 | Placebo
Number analyzed (Participants) | 44 | 43
Composite T-score | 0.8 [-1.0 to 2.6] | -0.2 [-2.0 to 1.5]
Statistical Analysis 1: Comparison: MK0249 vs Placebo; Test type: Superiority or Other; p = 0.736, constrained Logitudinal Data Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]

5. Other Pre Specified Outcome: Pre-randomization Baseline: Total Cognitive Score on the Brief Assessment of Cognition in Schizophrenia (BACS) Battery.
Description: Pre-randomization baseline values for all treatment sequences are equal because
  the constrained longitudinal data analysis (cLDA) model was used
  (Liang and Zeger, 2000, Sankhya: The Indian Journal of Statistics, Series B 62, 134-148).
Time Frame: Pre-randomization Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Composite T-score
Arm/Group | MK0249 | Placebo
Number analyzed (Participants) | 47 | 46
Composite T-score | 40.5 (0.98) | 40.5 (0.98)

6. Other Pre Specified Outcome: Pre-randomization Baseline: Attention/Processing Speed Composite Score
Description: as for outcome 5
Time Frame: Pre-randomization Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Composite T-score
Arm/Group | MK0249 | Placebo
Number analyzed (Participants) | 45 | 45
Composite T-score | 47.8 (0.73) | 47.8 (0.73)

7. Other Pre Specified Outcome: Pre-randomization Baseline: Episodic Memory Composite Score
Description: as for outcome 5
Time Frame: Pre-randomization Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Composite T-score
Arm/Group | MK0249 | Placebo
Number analyzed (Participants) | 47 | 45
Composite T-score | 43.9 (1.16) | 43.9 (1.16)

8. Other Pre Specified Outcome: Pre-randomization Baseline: Working Memory Composite Score
Description: as for outcome 5
Time Frame: Pre-randomization Baseline
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Composite T-score
Arm/Group | MK0249 | Placebo
Number analyzed (Participants) | 44 | 43
Composite T-score | 43.5 (0.98) | 43.5 (0.98)

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events (AEs) from visit 2 (V2) (Day -7): Neuropsych Testing through visit 11 (V11) (Day 77): 2-week Follow-Up.
Description: Abnormal Involuntary Movement Scale (AIMS), Simpson-Angus Scale (SAS), and Barnes Akathisia Rating Scale (BARS) were administered at visit 1 (V1), visit 6 (V6), and visit 10 (V10) to help assess for certain AEs.
Arm/Group | MK0249 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/52 | 0/51
Other Adverse Events (participants affected / at risk) | 20/52 | 15/51
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | MK0249 (N=52) | Placebo (N=51)
nausea (Gastrointestinal disorders) | 4 | 3
irritability (General disorders) | 0 | 3
nasopharyngitis (Infections and infestations) | 1 | 2
alanine aminotransferase increased (Investigations) | 1 | 2/48
aspartate aminotransferase increased (Investigations) | 0 | 2/48
blood creatine phosphokinase increased (Investigations) | 1 | 1/48
blood creatinine increased (Investigations) | 0 | 1/48
blood urea increased (Investigations) | 0 | 1/48
eosinophil count increased (Investigations) | 0 | 1/48
lymphocyte count increased (Investigations) | 0 | 1/48
neutrophil count decreased (Investigations) | 0 | 1/48
platelet count increased (Investigations) | 1 | 1/48
white blood cell count increased (Investigations) | 1 | 2/48
pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
headache (Nervous system disorders) | 6 | 2
anxiety (Psychiatric disorders) | 5 | 2
insomnia (Psychiatric disorders) | 7 | 4
middle insomnia (Psychiatric disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.